CLINICAL TRIAL: NCT03453398
Title: Effects of Shift Work on Health: Assessment of Sleep Quality, Motor Control and Cardiovascular Risk.
Brief Title: Effects of Shift Work on Nurse Staff Health
Acronym: Turnisti
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Turnisti
Record Dates: First submitted 2018-02-07; First posted 2018-03-05 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Shift Work Type Circadian Rhythm Sleep Disorder; Chronobiology Disorders; Mood Swing; Physical Activity; Cardiovascular Diseases
Keywords: Chronotype; Shift work; Health status
MeSH Terms: conditions — Chronobiology Disorders; Motor Activity; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: Participants are divided in three different groups on the bases of their actual shift work modalities. Thus no allocation process is possible within this project.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): Shifts over 24-hours, shift cycle of 5 days (morning, afternoon, night, night off, rest).
  Interventions: Other: Shifts working hours with different schedules
- Group 2 (Experimental): Shifts over 24-hours, shift cycle of 10 days (morning, morning, afternoon, afternoon, rest, night, night, night off, rest, rest).
  Interventions: Other: Shifts working hours with different schedules
- Group 3 (Active Comparator): Only diurnal shifts, shift cycle of 5 days (morning, afternoon, morning, afternoon, morning, rest, rest).
  Interventions: Other: Shifts working hours with different schedules

INTERVENTIONS:
Other: Shifts working hours with different schedules — Workers in Group 1, 2, and 3 will undergo three different shift work modalities presenting different schedules.
  Importantly, as an inclusion criteria, workers have to be involved in the same shift modality for at least one year at the time at the beginning of the study.

SUMMARY:
Shift work deeply impacts on temporal organization leading to a circadian desynchronization, which translates into a worsening of the sleep quality and work ability during waking hours. Furthermore, also the fine motor control skills and the subjective mood profile could undergo modifications in relation to the acquired sleep debt. The misalignment between working time and physiological/behavioral functions could have negative influences on the levels of spontaneous daily activity, with possible alteration of the activity-rest rhythm of the worker, especially in clinics.

In relation to the participants' chronotype, the aim of this project will be to evaluate the effect of irregular working hours (shift work) on (i) the sleep quality, (ii) the circadian rhythm of activity levels and, (iii) the motor control. These assessments will help to identify the shift type with less impact on the health status in a nurse cohort.

DETAILED DESCRIPTION:
Shift work can exert numerous effects on the temporal and behavioral organization of the individuals. Working hours of shift workers, which are outside the normal daily social program, lead to a circadian desynchronization due to a temporary misalignment between working time and physiological and behavioral functions, similarly to what is observed in the jet lag syndrome. This may lead to deterioration in the sleep quality, reduction in the working ability during waking hours, with sleepiness and a reduction in the vigilance state.

Over the years, the impact of shift work has involved many areas and its effects have been investigated at the cardiovascular (coronary artery disease, hypertension), metabolic (diabetes and obesity) and immunological level. Several investigations provided evidence of the shift work-induced negative results on health, including carcinogenic effects. Consequently, the scientific community paid to these problems great attention.

In analyzing the health effects of shift work, the chronotype of the workers, or their circadian typology, is very important. In fact, the circadian rhythms represent a dimension of the human personality that should not be underestimated. The human being has a temporal organization, determined by the interaction of endogenous and environmental factors, and organizes most of the biological and behavioral activities according to a twenty-four hour period and in sync with the light-dark cycle. It is not worthy to mention that the biological rhythms in humans present interindividual differences that determine precisely the chronotype, which is the tendency to express preferences toward morning or evening activities. Within the population, it is possible to recognize subjects that can be traced to three circadian types: (i) morning-types subjects (M-Types) that tend to be more active and efficient in the first part of the day, (ii) evening-types subjects (E-Types) who find it difficult to get up in the morning and require more time to reach the optimal level of physical and mental efficiency, and (iii) intermediate subjects (Neither-Types, N-Types) that present intermediate characteristics between the previous two.

Previous studies suggested that the eveningness could determine an easier adaptability to the changes determined by shift work. However, the role of the chronotype on this aspect is yet to be related to the type of shift: on one side, the E-Types tend to have more sleep disorders induced by a diurnal working shift. On the other side, the M-Types tend to adapt worst to a night working shift. In any case, shift work determines a growing sleep debt that can have a not negligible impact on the wellbeing and health of the individual.

The association between shift work and cardiovascular risk is very interesting. Sleep at night, in fact, can have important effects on blood pressure. Some studies have shown that a good sleep quality may have potential effects in the prevention of hypertension. Arterial pressure decreases by an average of 10-20% during nighttime hours, so sleep debt could lead to higher average blood pressure over the course of twenty-four hours. In addition, by modifying the circadian rhythms, the shift may lead to an alteration of the autonomic nervous system regulation with hypertensive consequences.

This project will focus on a particular category of shift workers, i.e., the nurse staff working in a hospital. Nurse staff has three different shift schedules: (i) shift changes every day (the first day from 7.00 to 14.00, the second day from 14.00 to 21.00, the third day from 21.00 to 7.00, the fourth day night off and, the fifth day rest), with a "shift cycle" duration of 5 days; (ii) shift changes every two days (first and second day from 7.00 to 14.00, third and fourth day from 14.00 to 21.00, fifth day rest, sixth and seventh day from 21.00 to 7.00, eighth day night off and ninth and tenth day rest), with a shift cycle of 10 days; and (iii) only diurnal shifts (first day from 7.00 to 14.00 and the second day from 14.00 to 21.00), with 2 days of rest every 5 work days.

To this purpose, the aim of this project will be to identify the type of shift work schedule with less impact on the state of health of the hospital staff by evaluating the effect of different shift work schedules on the quality of sleep, on the circadian rhythm of activity levels and on motor control, in relation to the participants' chronotype.

ELIGIBILITY:
Inclusion Criteria:

* Work shift continuity in a specific group of at least one year.

Exclusion Criteria:

* Presence of cardiovascular, endocrine or metabolic diseases;
* Presence of neurological or musculoskeletal impairments at finger flexors muscles level;
* Pharmacological therapies in place that can affect the heart rate and the sleep quality;
* Self-declaration of pregnancy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2018-01-23 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-01-15 (Actual)

PRIMARY OUTCOMES:
Sleep Efficiency (SE) | 8 days
  Percentage of time spent in bed with actual sleep
Sleep Latency (SL) | 8 days
  period of time between bed and sleep
Movement and Fragmentation Index (MFI) | 8 days
  Percentage of time spent moving indicative of the fragmentation of sleep
Immobile Time (IT) | 8 days
  total time spent without movement, between sleep from start to sleep
Assumed Sleep (AS) | 8 days
  Difference between beginning and end of sleep

SECONDARY OUTCOMES:
Profile of Mood States (POMS) | Baseline and 8 days
  Questionnaire for the determination of the mood profile
Finger flexor muscles maximum voluntary contraction (MVC) | Baseline and 8 days
  Evaluation of the maximum isometric force output of the finger flexors muscles
Force coefficient of variation (CV) | Baseline and 8 days
  Ratio between the standard deviation of the force signal during the plateau phase and the mean of the force signal (index of muscle contraction stability)
Distance of the force signal (DF) | Baseline and 8 days
  distance of the force signal with respect to the target (index of force accuracy )
Surface electromyography (sEMG) root mean square (RMS) of finger flexor muscles | Baseline and 8 days
  Index of muscle activation reflecting the number of recruited motor units during contraction
Surface electromyography (sEMG) mean frequency (MF) of finger flexor muscles | Baseline and 8 days
  Index reflecting the mean rate of activation of the recruited motor units during contraction
Hearth Rate Variability (HRV) | Baseline and 8 days
  Quantification of the sympatho-vagal balance

OTHER OUTCOMES:
Horne-Ostberg Morningness-Eveningness Questionnaire (MEQ) | Baseline
  Questionnaire for chronotype determination.The MEQ has 19 items, and the answer options include using a visual analog scale and choosing between four or five options. Participants are classified as Morning-types (scores between 59 and 86), Neither-types (scores between 42 and 58), and Evening-types (scores between 16 and 41).
International Physical Activity Questionnaire (IPAQ) | Baseline
  Questionnaire for the assessment of the level of physical activity. The number of days and minutes in a week dedicated at walking or in moderate or heavy physical activities are converted in metabolic equivalent units (METs). The sum of the METs identifies the level of physical activity: METs < 700 = inactive; METs from 700 to 2519 = adequately active; METs > 2519 highly active.
QRISK2-2017 questionnaire | Baseline
  Questionnaire for cardiovascular risk assessment. The questionnaire provides a score (in percentage) of the risk of having a heart attack or stroke within the next 10 years. Score ranges from 0.1% (lowest risk) and 100% (maximum risk).

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Esposito, MD, Principal Investigator — University of Milan
Locations (1):
- IRCCS Istituto Ortopedico Galeazzi, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: Yes
Anonymous individual participant data for all primary and secondary outcome measures will be made available
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available within 6 months from the end of the study.
Access Criteria: Data access request will be reviewed by the principal investigator and co-investigators.
  Requestors will be required to sign a Data Access Agreement.

REFERENCES:
- [Background] Adan A, Archer SN, Hidalgo MP, Di Milia L, Natale V, Randler C. Circadian typology: a comprehensive review. Chronobiol Int. 2012 Nov;29(9):1153-75. doi: 10.3109/07420528.2012.719971. Epub 2012 Sep 24. PMID 23004349
- [Background] Akerstedt T. Shift work and disturbed sleep/wakefulness. Sleep Med Rev. 1998 May;2(2):117-28. doi: 10.1016/s1087-0792(98)90004-1. PMID 15310506
- [Background] Boivin DB, Tremblay GM, James FO. Working on atypical schedules. Sleep Med. 2007 Sep;8(6):578-89. doi: 10.1016/j.sleep.2007.03.015. Epub 2007 May 3. PMID 17481949
- [Background] Costa G, Anelli MM, Castellini G, Fustinoni S, Neri L. Stress and sleep in nurses employed in "3 x 8" and "2 x 12" fast rotating shift schedules. Chronobiol Int. 2014 Dec;31(10):1169-78. doi: 10.3109/07420528.2014.957309. Epub 2014 Sep 12. PMID 25216205
- [Background] Guo Y, Liu Y, Huang X, Rong Y, He M, Wang Y, Yuan J, Wu T, Chen W. The effects of shift work on sleeping quality, hypertension and diabetes in retired workers. PLoS One. 2013 Aug 16;8(8):e71107. doi: 10.1371/journal.pone.0071107. eCollection 2013. PMID 23976988
- [Background] Halberg F, Carandente F, Cornelissen G, Katinas GS. [Glossary of chronobiology (author's transl)]. Chronobiologia. 1977;4 Suppl 1:1-189. No abstract available. Italian. PMID 352650
- [Background] Harma M. Individual differences in tolerance to shiftwork: a review. Ergonomics. 1993 Jan-Mar;36(1-3):101-9. doi: 10.1080/00140139308967860. PMID 8440205
- [Background] Hippisley-Cox J, Coupland C, Robson J, Brindle P. Derivation, validation, and evaluation of a new QRISK model to estimate lifetime risk of cardiovascular disease: cohort study using QResearch database. BMJ. 2010 Dec 9;341:c6624. doi: 10.1136/bmj.c6624. PMID 21148212
- [Background] Hippisley-Cox J, Coupland C, Vinogradova Y, Robson J, Minhas R, Sheikh A, Brindle P. Predicting cardiovascular risk in England and Wales: prospective derivation and validation of QRISK2. BMJ. 2008 Jun 28;336(7659):1475-82. doi: 10.1136/bmj.39609.449676.25. Epub 2008 Jun 23. PMID 18573856
- [Background] Horne JA, Ostberg O. A self-assessment questionnaire to determine morningness-eveningness in human circadian rhythms. Int J Chronobiol. 1976;4(2):97-110. PMID 1027738
- [Background] Juda M, Vetter C, Roenneberg T. Chronotype modulates sleep duration, sleep quality, and social jet lag in shift-workers. J Biol Rhythms. 2013 Apr;28(2):141-51. doi: 10.1177/0748730412475042. PMID 23606613
- [Background] Martin JS, Laberge L, Sasseville A, Berube M, Alain S, Houle J, Hebert M. Day and night shift schedules are associated with lower sleep quality in Evening-types. Chronobiol Int. 2015 Jun;32(5):627-36. doi: 10.3109/07420528.2015.1033425. Epub 2015 Jun 2. PMID 26035480
- [Background] Montaruli A, Galasso L, Caumo A, Cè E, Pesenti C, Roveda E, Esposito F. (2017). The circadian typology: the role of physical activity and melatonin. Sport Sciences for Health 1-8, 2017
- [Background] Montaruli A, Galasso L, Carandente F, Vitale JA, Roveda E, Caumo A. If the Morning-Evening Questionnaire (MEQ) is able to predict the actigraphy-based acrophase, how does its reduced, five-item version (rMEQ) perform? Chronobiol Int. 2017;34(4):443-444. doi: 10.1080/07420528.2017.1306708. No abstract available. PMID 28426388
- [Background] Nelson W, Tong YL, Lee JK, Halberg F. Methods for cosinor-rhythmometry. Chronobiologia. 1979 Oct-Dec;6(4):305-23. No abstract available. PMID 548245
- [Background] Newey CA, Hood BM. Determinants of shift-work adjustment for nursing staff: the critical experience of partners. J Prof Nurs. 2004 May-Jun;20(3):187-95. doi: 10.1016/j.profnurs.2004.04.007. PMID 15211428
- [Background] Rajaratnam SM, Arendt J. Health in a 24-h society. Lancet. 2001 Sep 22;358(9286):999-1005. doi: 10.1016/S0140-6736(01)06108-6. PMID 11583769
- [Background] Roveda E, Vitale JA, Bruno E, Montaruli A, Pasanisi P, Villarini A, Gargano G, Galasso L, Berrino F, Caumo A, Carandente F. Protective Effect of Aerobic Physical Activity on Sleep Behavior in Breast Cancer Survivors. Integr Cancer Ther. 2017 Mar;16(1):21-31. doi: 10.1177/1534735416651719. Epub 2016 Jun 1. PMID 27252076
- [Background] Roveda E, Vitale J, Montaruli A, Galasso L, Carandente F, Caumo A. Predicting the actigraphy-based acrophase using the Morningness-Eveningness Questionnaire (MEQ) in college students of North Italy. Chronobiol Int. 2017;34(5):551-562. doi: 10.1080/07420528.2016.1276928. Epub 2017 Feb 21. PMID 28276851
- [Background] Saksvik IB, Bjorvatn B, Hetland H, Sandal GM, Pallesen S. Individual differences in tolerance to shift work--a systematic review. Sleep Med Rev. 2011 Aug;15(4):221-35. doi: 10.1016/j.smrv.2010.07.002. Epub 2010 Sep 20. PMID 20851006
- [Background] Schernhammer ES, Laden F, Speizer FE, Willett WC, Hunter DJ, Kawachi I, Colditz GA. Rotating night shifts and risk of breast cancer in women participating in the nurses' health study. J Natl Cancer Inst. 2001 Oct 17;93(20):1563-8. doi: 10.1093/jnci/93.20.1563. PMID 11604480
- [Background] Munakata M, Ichi S, Nunokawa T, Saito Y, Ito N, Fukudo S, Yoshinaga K. Influence of night shift work on psychologic state and cardiovascular and neuroendocrine responses in healthy nurses. Hypertens Res. 2001 Jan;24(1):25-31. doi: 10.1291/hypres.24.25. PMID 11213026
- [Derived] Galasso L, Mule A, Castelli L, Ce E, Condemi V, Banfi G, Roveda E, Montaruli A, Esposito F. Effects of Shift Work in a Sample of Italian Nurses: Analysis of Rest-Activity Circadian Rhythm. Int J Environ Res Public Health. 2021 Aug 8;18(16):8378. doi: 10.3390/ijerph18168378. PMID 34444128

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-10-02): https://cdn.clinicaltrials.gov/large-docs/98/NCT03453398/Prot_SAP_000.pdf
  • Informed Consent Form (2017-12-19): https://cdn.clinicaltrials.gov/large-docs/98/NCT03453398/ICF_001.pdf